CLINICAL TRIAL: NCT07008833
Title: Randomized, Non-inferiority Study Comparing Radiochemotherapy Versus Radical Cystectomy in Patients With Muscle-invasive Bladder Cancer
Brief Title: Radical CystEctomy or RaDio-chEMotherapy as Preferred Treatment for invasivE blaDder Cancer
Acronym: REDEMPTED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002/2024; 01245.011245/2023-57 (Other: Parliamentary Amendment Ministry of Science, Technology, Innovation and Communications)
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Bladder cancer; Radiochemotherapy; Radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Chemoradiotherapy; Cystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical outcomes will be independently ascertained by a Clinical Events Committee, whose members will not be aware of the study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Maximum TURBT + neoadjuvant chemotherapy with cisplatin + radiotherapy
  Interventions: Procedure: Radiochemotherapy
- Arm 2 (Other): TURBT + neoadjuvant chemotherapy with cisplatin + radical cystectomy, bilateral pelvic lymphadenectomy + reconstruction
  Interventions: Procedure: Radical cystectomy

INTERVENTIONS:
Procedure: Radiochemotherapy — Maximum TURBT will be followed by neoadjuvant chemotherapy with cisplatin at a dose of 35 mg/m². After 2-6 weeks of neoadjuvant chemotherapy, patients will receive radiotherapy for 4 weeks, with concomitant cisplatin at a dose of 40 mg/m² weekly.
  Arms: Arm 1
Procedure: Radical cystectomy — TURBT will be followed by neoadjuvant chemotherapy with cisplatin at a dose of 35 mg/m², followed by radical cystectomy, bilateral pelvic lymphadenectomy, and reconstruction with either a Bricker procedure or a neobladder.
  Arms: Arm 2

SUMMARY:
Your text is mostly clear and well-structured. Here's a slightly polished version for improved clarity and flow:

This is a randomized, non-inferiority study comparing radiochemotherapy to radical cystectomy in patients with muscle-invasive bladder cancer. The primary outcome is the evaluation of the non-inferiority of metastasis-free survival between the two treatments.

The study population includes individuals of both sexes, aged 18 years and older, diagnosed with pure or predominant urothelial carcinoma. Participants will be randomized in a 1:1 ratio, with Arm 1 receiving maximal TURBT followed by neoadjuvant chemotherapy and radiotherapy, and Arm 2 receiving TURBT followed by neoadjuvant chemotherapy with cisplatin, followed by radical cystectomy and bilateral pelvic lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Pure or predominant urothelial carcinoma (including other histologic subtypes, with the exception of small cell carcinoma, as a minority component).
3. Performance status of 0 to 1, according to the Eastern Cooperative Oncology Group (ECOG) criteria.
4. Life expectancy of ≥ 3 months.
5. Histologically confirmed T2, T3, or T4a stage bladder cancer (pure or predominant urothelial carcinoma) cN0 or cN1 or cN2 (if lymph nodes within the surgical and radiation fields and size ≤ 2 cm).
6. Patients who are candidates for neoadjuvant cisplatin and have undergone TURBT (preferably maximal) prior to treatment.
7. Adequate bladder function (defined as the ability to store and void urine effectively, without symptoms of dysfunction or incontinence).
8. Neutrophil count ≥ 1500/mm³.
9. Platelet count ≥ 100,000/mm³.
10. Hemoglobin count > 10 g/dL.
11. Glomerular filtration rate greater than 40 mL/min.
12. Serum bilirubin < 1.5 times the upper limit of the normal reference range and SGOT and SGPT < 1.5 times the upper limit of the normal reference range.
13. Absence of comorbidities that contraindicate treatment.
14. Capable of giving signed and dated informed consent prior to any mandatory study-specific procedures, sampling, and analyses, which includes compliance with the requirements and restrictions listed in the informed consent form and study protocol.
15. For inclusion in i) optional exploratory genetic research and ii) optional biomarker research, patients must meet the following criteria:

    * Provide informed consent for genetic research prior to sample collection.
    * Provide informed consent for biomarker research prior to sample collection.
    * If a patient declines to participate in optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Exclusion Criteria:

1. Presence of multiple primary tumors or multiple foci of carcinoma in situ (CIS) (including in the upper tract) that are not candidates for bladder preservation with radiochemotherapy (definition at the discretion of the investigator).
2. Age > 80 years.
3. Pure adenocarcinoma or pure squamous carcinoma or pure small cell or large cell neuroendocrine carcinoma, micropapillary, sarcomatoid or nested.
4. Metastatic or unresectable disease.
5. Sensory neuropathy Grade ≥ 2.
6. Hearing impairment Grade ≥ 2.
7. Having a known additional malignancy that has progressed or required active treatment in the last 5 years, except superficial bladder cancer and/or carcinoma in situ, basal cell carcinoma of the skin or carcinoma in situ of the cervix.
8. Clinically significant cardiovascular disease - functional class III-IV according to the New York Heart Association (NYHA) Classification of heart failure.
9. Patients considered to be at high medical risk due to severe and uncontrolled disease, active or non-malignant systemic disease, and severe or potentially severe infection that may affect response to treatment or increase the risk of adverse events.
10. Immunocompromised patients.
11. Inflammatory bowel disease.
12. Patients with known active hepatitis (i.e., hepatitis B or C).
13. Patients receiving any prior systemic chemotherapy in the last 5 years for other tumors and at any time for muscle-invasive bladder cancer.
14. Patients who have received prior systemic immunotherapy at any time, either in the setting of non-muscle-invasive bladder cancer or in treatment for other types of cancer.
15. Prior pelvic radiotherapy.
16. Patients, male or female, who do not agree to use an effective method of contraception throughout treatment and until 6 months after discontinuation of treatment.
17. Women who are pregnant or currently breastfeeding. 18. The investigator's judgment that the patient should not participate in the study if the patient is unlikely to comply with the procedures, restrictions, and requirements.

19. Prior Randomization to the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | The time from the start of treatment until detection of 230 metastases in other organs or tissues outside the bladder (including pelvic lymph nodes).or until death from any cause of the patient, estimated to be up to 8 years
  The primary outcome is the assessment of the non-inferiority of metastasis-free survival between radiochemotherapy and radical cystectomy.

SECONDARY OUTCOMES:
Overall survival | The duration from treatment initiation until the study accrues 230 patients with a primary event, or 6 years of follow-up
  Overall survival of radiochemotherapy versus radical cystectomy.
Muscle-invasive bladder cancer-free survival | The duration from treatment initiation until the study accrues 230 patients with a primary event, or 6 years of follow-up
Incidence of tumors in the upper tract (in both arms) | The duration from treatment initiation until the study accrues 230 patients with a primary event, or 6 years of follow-up
  The proportion of patients who develop new tumors in the upper urinary tract in 6 years
Adverse Events assessment | The duration from treatment initiation until the study accrues 230 patients with a primary event, or 6 years of follow-up
  All adverse events will be collected and classified according to CTCAE v5.0. The protocol defines the following adverse events of special interest for the Radical Cystectomy group: surgical (infections, bleeding, organ injury, thromboembolism), postoperative (fistula, stricture, hernia, delayed healing), and long-term complications (renal insufficiency, GI disorders, sexual dysfunction, body image issues). And Chemoradiotherapy group: acute effects (cystitis, proctitis, enteritis, nausea, vomiting) and severe toxicities (hematologic toxicity, grade 3-4 diarrhea, skin toxicity).
Quality of Life assessment | The duration from treatment initiation until the study accrues 230 patients with a primary event, or 6 years of follow-up
  Assessment of the perception of patients with bladder cancer about their general well-being, including symptoms of the disease, impact of treatment, psychological and emotional aspects, and the ability to perform physical and social activities, measured through the EORTC QLQ-BLM30 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Brazilian Clinical Research Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided